CLINICAL TRIAL: NCT03650790
Title: Diyarbakir Women's and Children's Diseases Hospital
Brief Title: C1q/TNF-related Protein 9 (CTRP 9) Level in Preeclamptic Obese and Non-obese Pregnancies
Acronym: CTRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diyarbakir Women's and Children's Diseases Hospital (Other)
Responsible Party: Principal Investigator, Şerif AKSİN, specialist doctor, Diyarbakir Women's and Children's Diseases Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DiyarbakirWCDH
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Pre-Eclampsia; Obesity; Endocrine
Keywords: CTRP; Adipocytokines; pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia; Obesity | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: 40 obese preeclamptic pregnant women 40 non-obese preeclamptic pregnant women 40 normal pregnant women
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- preeclamptic obese pregnancy (Active Comparator): CTRP 9 level will be assessed by 40 obese preeclamptic gestational ELISA methods that meet the latest ACOG criteria.
  Interventions: Diagnostic Test: Blood test
- preeclamptic non-obese pregnancy (Active Comparator): CTRP 9 level will be assessed by 40 non-obese preeclamptic gestational ELISA methods that meet the latest ACOG criteria.
  Interventions: Diagnostic Test: Blood test
- normal pregnancy (Active Comparator): CTRP 9 level will be assessed by 40 normal gestational ELISA methods
  Interventions: Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Blood test — For serum analysis, approximately 2 cc antecubital vein venous blood serum will be taken from each patient to be studied for CTRP9 Level analysis. Adult blood will be centrifuged at 4000 rpm for 10 minutes to separate greenhouses. The obtained serum samples will be stored at -80 ° C until analysis.

SUMMARY:
The complement C1q tumor necrosis factor-associated protein-9 (CTRP-9), which is responsible for regulating cardiovascular and metabolic functions, increases vascular relaxation by pathway dependent on AMPK / endothelial nitric oxide synthesis (eNOS). The aim of this study was to investigate CTRP-9 levels in pregnant women with preeclampsia.

DETAILED DESCRIPTION:
The most important reason for the development of preeclampsia is the problem of trophoblastinvasion and consequent formation and development of placenta is not healthy

Cytokines are regulatory molecules that have effects on cell functions.Cytokines are molecules that also regulate endothelial functions. Placenta formation and widespread endothelial damage are under the influence of cytokines.

Therefore, there may be important links between impairment or imbalance in cytokine release and function and the formation of preeclampsia.Nitric oxide (NO) is a biologic enzyme that is synthesized by nitric oxide synthase (NOS) from the amino acid of L-arginine and exists in all mammals.

e(NOS) is the three isoforms of NO. It is known that NO is a major vasodilator of pregnancy, inhibiting platelet and leukocyte aggregation.There was a decrease in NO levels in preeclamptic patients.

The CqP / TNF Binding Protein (CTRP) family consists of 15 members, and is synthesized in many organs outside the body of fat.CTRP9 is predominantly excreted in fat tissue, and levels in circulation are reduced in patients with diabetes and obesity.Many studies have shown that CTRP9 exerts beneficial effects on metabolic and cardiovascular homeostasis.

CTRP9 increases vascular relaxation in the AMPK / endothelial nitric oxide synthase (eNOS) dependent pathway. CTRP9 has also been reported to reduce inflammatory responses in endothelial cells via the AMPK-dependent pathway.

Vasorelaxation due to CTRP9 is endothelium-dependent and NO-mediated. CTRP9, directly acting on smooth muscle, is indirectly or indirectly associated with NO production in the vascular endothelial layer by stimulating vasorelaxial molecular production by endothelial cells.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are ages 15-40
* BMI ≥35 kg/m2 and BMI<25 KG/m2 pregnants
* The clinical diagnosis of preeclampsia will follow the current criteria outlined by ACOG 10
* > 20 th weeks of pregnancy

Exclusion Criteria:

* A previously known chronic metabolic disease (diabetes, pregestational dyslipidemia, hypertension,)
* collagen vascular diseases,
* inflammatory bowel disease
* chronic inflammatory conditions,

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
CTRP 9 level in preeclamptic pregnancies | 3 months
  Blood samples were taken from patients with preeclampsia. The diagnosis was made when the arterial blood pressure was above 140/90 mm / Hg within 6 hours and was accompanied by proteinuria (> 300 milligrams in a sample) with high blood pressure and number of patients with proteinuria (ACOG criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Şerif Aksin, specialist, Principal Investigator — Diyarbakir Women's and Children's Diseases Hospital
Locations (1):
- Diyarbakır Women's and Children's Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Preeclampsia relationship of adipocytokines — https://www.ncbi.nlm.nih.gov/pubmed/21836066
- See also: Relation to CTRP 9 vasodilatation — https://www.ncbi.nlm.nih.gov/pubmed/30103635